CLINICAL TRIAL: NCT00473746
Title: Phase I/II Open Label Dose Escalation Study of the 17α-Hydroxylase/ C17,20-Lyase Inhibitor, Abiraterone Acetate in Hormone Refractory Prostate Cancer
Brief Title: Abiraterone Acetate Dose-Escalation Study in Hormone Refractory Prostate Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR016969; COU-AA-002 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2007-05-11; First posted 2007-05-15 (Estimated); Results first posted 2014-04-29 (Estimated); Last update posted 2014-04-29 (Estimated); Status verified 2014-03

CONDITIONS: Prostate Neoplasms
Keywords: Prostate neoplasms; Hormone refractory prostate cancer; Abiraterone acetate; CB7630
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Abiraterone Acetate; Prednisone; Prednisolone; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Phase I Dose Escalation (Experimental)
  Interventions: Drug: Abiraterone acetate
- Phase II Dose Treatment (Experimental)
  Interventions: Drug: Abiraterone acetate; Drug: prednisone/prednisolone or dexamethasone

INTERVENTIONS:
Drug: Abiraterone acetate — The first cohort was a abiraterone acetate 250 mg/day orally (by mouth), once daily for 28-day treatment periods , if no dose limiting toxicity (DLT) was documented at this dose, the dose will be escalated to next dose levels 500, 750, and 1000 mg/day. The dose escalation will continue to a maximum of 1000mg/day until Maximum Tolerated Dose (MTD) and a recommended Phase II dose was established.
  Arms: Phase I Dose Escalation
Drug: Abiraterone acetate — Abiraterone acetate 1000 mg daily under fasted conditions upto 10 cycles of therapy.
  Arms: Phase II Dose Treatment
Drug: prednisone/prednisolone or dexamethasone — prednisone/prednisolone (5 mg twice daily) or dexamethasone (0.5 mg once daily) concurrent with abiraterone acetate
  Arms: Phase II Dose Treatment

SUMMARY:
The purpose of this study is to evaluate the safety, pharmacokinetics, pharmacodynamics, and anti-tumor activities of abiraterone acetate (also referred to as CB7630) in patients with hormone refractory prostate cancer (HRPC).

DETAILED DESCRIPTION:
This is an open-label (identity of assigned study drug will be known) study to evaluate the safety, pharmacokinetics (study of what the body does to a drug), pharmacodynamics (study of what a drug does to the body), and anti-tumor activities of abiraterone acetate (also known as CB7630) in patients with HRPC. The study will be conducted in 2 phases (Phase 1 and Phase 2). In the first part of the study (Phase 1), the maximum tolerated dose (MTD) of abiraterone acetate will be determined for use in the second part of the study (Phase 2) where the number of patients who achieve at least a 50% decrease in prostate specific antigen (PSA) during treatment with abiraterone acetate will be assessed (MTD from Phase 1). Abiraterone acetate will be taken orally (by mouth) in fed and fasted patients once daily. Doses of abiraterone acetate (starting at 250 mg up to a maximum of 2000 mg) will be taken for 28-day treatment periods to determine the MTD. Patients will take MTD of abiraterone acetate for up to twelve 28 day cycles (12 months; patients will be given the option of staying on abiraterone acetate treatment if they are deriving benefit). In Phase 2, prednisone or dexamethasone will be administered concurrently with abiraterone acetate. Serial pharmacokinetic and pharmacodynamic samples will be collected and safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

Phase 1

* Histologically confirmed adenocarcinoma of the prostate
* No prior therapy with chemotherapy for prostate cancer
* Ongoing gonadal androgen deprivation therapy with luteinizing hormone-releasing hormone (LHRH) analogues or orchiectomy
* Testosterone <50 ng/dL
* Progressive disease after androgen deprivation
* The presence of objective metastatic disease is NOT required for study eligibility
* Demonstrate disease progression after antiandrogen withdrawal
* Eastern Cooperative Oncology Group (ECOG) performance status score = 0-1
* Laboratory values within protocol-defined parameters
* Systolic blood pressure <160 mmHg and diastolic blood pressure <110mmHg documented on at least 3 different days
* Baseline adrenocorticotropic hormone (ACTH) stimulation test demonstrating a peak cortisol >18 µg/dL
* Agrees to protocol-defined use of effective contraception
* Life expectancy of >=12 weeks

Phase 2

* Same as Phase 1 criteria with addition of following criteria
* Neoadjuvant or adjuvant chemotherapy is only allowed if the last dose is >1 year from Cycle 1 Day 1
* Target or non-target abnormalities must be present either on screening bone scan, computed tomography or magnetic resonance imaging
* No prior treatment with ketoconazole for the management of androgen independent prostate cancer

Exclusion Criteria:

Phase 1

* Therapy with other hormonal therapy, including any dose of megestrol acetate (Megace), finasteride (Proscar), dutasteride (Avodart) any herbal product known to decrease prostate specific antigen (PSA) levels (eg, saw palmetto and PC-SPES), or any systemic corticosteroid within 4 weeks prior to first dose of study drug
* Initiation of bisphosphonate therapy within 4 weeks prior to first dose of study drug
* Therapy with supplements or complementary medicines/botanicals within 4 weeks of first dose of study drug, except for any combination of the following: conventional multivitamin supplements, selenium, lycopene, soy supplements
* Prior radiation therapy completed <4 weeks prior to enrollment
* Prior chemotherapy for hormone refractory prostate cancer
* Any currently active second malignancy, other than non-melanoma skin cancer
* Systolic blood pressure >=160 mmHg or diastolic blood pressure >=110 mmHg measured on at least 2 occasions
* NYHA Class III or IV congestive heart failure
* Myocardial infarction within the 6 months prior to the first dose of study drug
* Serious intercurrent infections or nonmalignant medical illnesses that are uncontrolled
* Active psychiatric illnesses/social situations that would limit compliance with protocol requirements
* Active or uncontrolled autoimmune disease that may require corticosteroid therapy during study

Phase 2

* Same as phase 1 with the following addition
* Abnormal electrocardiogram, including any finding which would interfere with assessment of intervals (patients with long QT syndrome, bundle branch blocks or hemiblocks are prohibited)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2006-06; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (3):
- United States (3):
  - San Francisco, California
  - Boston, Massachusetts
  - Houston, Texas

REFERENCES:
- [Derived] Aggarwal R, Harris A, Formaker C, Small EJ, Molina A, Griffin TW, Ryan CJ. Response to subsequent docetaxel in a patient cohort with metastatic castration-resistant prostate cancer after abiraterone acetate treatment. Clin Genitourin Cancer. 2014 Oct;12(5):e167-72. doi: 10.1016/j.clgc.2014.03.010. Epub 2014 Mar 28. PMID 24787968
- See also: NATIONAL CANCER INSTITUTE — http://www.cancer.gov/
- See also: PROSTATE CANCER — http://www.nlm.nih.gov/medlineplus/prostatecancer.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted between 10 July 2006 and 22 December 2012.
Pre-assignment Details: 66 participants participated in the study, including 33 participants enrolled in Phase 1 of the study, and 33 participants enrolled in Phase 2 of the study.
Groups:
- Phase 1 250 MG/DAY; Phase 1 500 MG/DAY; Phase 1 750 MG/DAY; Phase 1 1000 MG/DAY; Phase 2 1000 MG/DAY: Abiraterone acetate
Period: Period 1 (Phase 1)
Arm/Group | Phase 1 250 MG/DAY | Phase 1 500 MG/DAY | Phase 1 750 MG/DAY | Phase 1 1000 MG/DAY | Phase 2 1000 MG/DAY
Started | 6 | 9 | 6 | 12 | 0
Completed | 0 | 0 | 0 | 2 (Treatment ongoing) | 0
Not Completed | 6 | 9 | 6 | 10 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0
Not completed — Progressive Disease | 5 | 6 | 6 | 10 | 0
Not completed — Symptomatic Deterioration | 0 | 1 | 0 | 0 | 0
Not completed — Reason not specified | 0 | 1 | 0 | 0 | 0
Period: Period 2 (Phase 2)
Arm/Group | Phase 1 250 MG/DAY | Phase 1 500 MG/DAY | Phase 1 750 MG/DAY | Phase 1 1000 MG/DAY | Phase 2 1000 MG/DAY
Started | 0 | 0 | 0 | 0 | 33
Completed | 0 | 0 | 0 | 0 | 6
Not Completed | 0 | 0 | 0 | 0 | 27
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 3
Not completed — Death | 0 | 0 | 0 | 0 | 1
Not completed — Progressive Disease | 0 | 0 | 0 | 0 | 20
Not completed — Reason not specified | 0 | 0 | 0 | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase 1 250 MG/DAY | Phase 1 500 MG/DAY | Phase 1 750 MG/DAY | Phase 1 1000 MG/DAY | Phase 2 1000 MG/DAY | Total
Number analyzed (Participants) | 6 | 9 | 6 | 12 | 33 | 66
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.7 (6.19) | 67.6 (6.5) | 73.2 (8.18) | 72.9 (8.3) | 70.3 (8.51) | 70.3 (8.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0
  Male | 6 | 9 | 6 | 12 | 33 | 66
Region of Enrollment [Number; unit: participants]
  United States | 6 | 9 | 6 | 12 | 33 | 66

OUTCOME MEASURES:

1. Primary Outcome: Phase 1: Maximum Tolerated Dose (MTD) of Abiraterone Acetate
Description: The MTD is the highest dose of a drug or treatment that does not cause unacceptable side effects.
Time Frame: Up to Cycle 12
Population: Safety population included all enrolled participants who received any study drug. MTD of abiraterone acetate was not reached because the doses administered appear to be well tolerated with no Dose Limiting Toxicity (DLT) even at 1000 milligram per day (mg/day [recommended maximum dose for phase 1]) and 1000 mg/day was taken as test dose in phase 2.
Measure: Number; unit: mg/day
Groups:
- Phase I Dose Escalation: The first cohort was a abiraterone acetate 250 mg/day orally (by mouth), once daily for 28-day treatment periods , if no dose limiting toxicity (DLT) was documented at this dose, the dose will be escalated to next dose levels 500, 750, and 1000 mg/day. The dose escalation will continue to a maximum of 1000 mg/day until maximum tolerated dose (MTD) and a recommended Phase II dose was established.
Arm/Group | Phase I Dose Escalation
Number analyzed (Participants) | 33
mg/day | NA (0) — MTD of abiraterone acetate was not reached because the doses administered appear to be well tolerated with no Dose Limiting Toxicity (DLT) even at 1000 milligram per day.

2. Primary Outcome: Phase 2: Participants With Greater Than or Equal to 50 Percent Decline in Prostate Specific Antigen (PSA)
Description: Number of participants with greater than or equal to 50 percent decrease in PSA levels were assessed. PSA decline was evaluated according to (Prostate Specific Antigen Working Group) PSAWG criteria. Decrease in PSA levels represented improvement.
Time Frame: Up to 12 weeks from start of treatment
Population: Intent-to-treat (ITT) population included all participants who were enrolled into the study.
Measure: Number; unit: participants
Groups:
- Phase II Dose Treatment: Abiraterone acetate 1000 mg daily and concurrent prednisone/prednisolone (5 mg twice daily) or dexamethasone (0.5 mg once daily) under fasted conditions upto 10 cycles of therapy.
Arm/Group | Phase II Dose Treatment
Number analyzed (Participants) | 33
participants
  Confirmed | 26
  Not Confirmed | 2
  Total | 28

3. Secondary Outcome: Phase 1: Maximum Plasma Concentration (Cmax) of Abiraterone Acetate
Description: Blood samples for pharmacokinetic (PK) measurements was taken on Day -7 at hour 0 (predose), at hours 1, 2, 4, 6, 8, and 12 (postdose). On Day -6 at 24 hour (postdose) and Day -5 at 48 hour (postdose). On Days 1, 8, 15, 22 of Cycle 1 and Day 1 of Cycles 2 and 3 (Predose).
Time Frame: At hours 1, 2, 4, 6, 8, 12, 24 and 48 post dose and pre-dose on day 1, day 8, day 15 and day 22 cycle 1, day 1 cycle 2 and day 1 cycle 3.
Population: ITT population included all participants who were enrolled into the study.
Measure: Mean (Standard Deviation); unit: nanomoles per liter (nmol/L)
Groups:
- Phase I Dose Escalation (250mg): The first cohort was a abiraterone acetate 250 mg/day orally (by mouth), once daily for 28-day treatment periods.
- Phase I Dose Escalation (500mg): The second cohort was a abiraterone acetate 500 mg/day orally (by mouth), once daily for 28-day treatment periods.
- Phase I Dose Escalation (750mg): The third cohort was a abiraterone acetate 700 mg/day orally (by mouth), once daily for 28-day treatment periods.
- Phase I Dose Escalation (1000mg): The fourth cohort was a abiraterone acetate 1000 mg/day orally (by mouth), once daily for 28-day treatment periods.
Arm/Group | Phase I Dose Escalation (250mg) | Phase I Dose Escalation (500mg) | Phase I Dose Escalation (750mg) | Phase I Dose Escalation (1000mg)
Number analyzed (Participants) | 6 | 9 | 6 | 12
nanomoles per liter (nmol/L)
  Fasted | 283.000 (142.265) | 330.633 (204.889) | 289.533 (126.646) | 509.500 (366.452)
  Fed | 421.000 (75.809) | 676.000 (147.866) | 1552.000 (458.082) | 2194.250 (1096.914)

4. Secondary Outcome: Phase 1: Time to Reach the Maximum Plasma Concentration (Tmax) of Abiraterone Acetate
Description: as for outcome 3
Time Frame: as for outcome 3
Population: ITT population included all participants who were enrolled into the study.
Measure: Mean (Standard Deviation); unit: hour (hr)
Arm/Group | Phase I Dose Escalation (250mg) | Phase I Dose Escalation (500mg) | Phase I Dose Escalation (750mg) | Phase I Dose Escalation (1000mg)
Number analyzed (Participants) | 6 | 9 | 6 | 12
hour (hr)
  Fasted | 2.000 (0.000) | 1.500 (0.548) | 2.033 (0.058) | 1.833 (0.408)
  Fed | 2.044 (0.077) | 2.667 (1.155) | 2.000 (0.000) | 4.000 (0.000)

5. Secondary Outcome: Phase 1: Area Under the Plasma-Concentration-Time Curve From Time 0 to the Last Quantifiable Concentration (AUClast) of Abiraterone Acetate
Description: as for outcome 3
Time Frame: as for outcome 3
Population: ITT population included all participants who were enrolled into the study.
Measure: Mean (Standard Deviation); unit: hr*nmol/L
Arm/Group | Phase I Dose Escalation (250mg) | Phase I Dose Escalation (500mg) | Phase I Dose Escalation (750mg) | Phase I Dose Escalation (1000mg)
Number analyzed (Participants) | 6 | 9 | 6 | 12
hr*nmol/L
  Fasted | 1329.178 (699.977) | 1625.059 (930.364) | 1565.659 (661.289) | 3039.937 (1902.697)
  Fed | 1310.715 (311.041) | 3624.781 (1041.927) | 8920.790 (3060.457) | 13695.482 (5623.185)

6. Secondary Outcome: Phase 1: Area Under the Plasma-Concentration-time Curve From Time 0 to Infinite Time (AUCINF_obs) of Abiraterone Acetate
Description: as for outcome 3
Time Frame: as for outcome 3
Population: ITT population included all participants who were enrolled into the study.
Measure: Mean (Standard Deviation); unit: hr*nmol/L
Arm/Group | Phase I Dose Escalation (250mg) | Phase I Dose Escalation (500mg) | Phase I Dose Escalation (750mg) | Phase I Dose Escalation (1000mg)
Number analyzed (Participants) | 6 | 9 | 6 | 12
hr*nmol/L
  Fasted | 1411.268 (697.183) | 1781.374 (986.770) | 1665.454 (704.551) | 3478.385 (2012.176)
  Fed | 1386.939 (290.240) | 3839.804 (1080.853) | 9358.743 (3338.601) | 14404.387 (5971.041)

7. Secondary Outcome: Phase 1: Terminal Half-life (HL_Lambda_z) of Abiraterone Acetate
Description: as for outcome 3
Time Frame: as for outcome 3
Population: ITT population included all participants who were enrolled into the study.
Measure: Mean (Standard Deviation); unit: hour (hr)
Arm/Group | Phase I Dose Escalation (250mg) | Phase I Dose Escalation (500mg) | Phase I Dose Escalation (750mg) | Phase I Dose Escalation (1000mg)
Number analyzed (Participants) | 6 | 9 | 6 | 12
hour (hr)
  Fasted | 5.284 (1.676) | 10.591 (6.337) | 7.066 (3.431) | 14.361 (7.655)
  Fed | 5.125 (1.039) | 6.913 (5.720) | 7.939 (2.633) | 12.454 (1.218)

8. Secondary Outcome: Phase 1: Total Body Clearance (Cl_F_obs) of Abiraterone Acetate
Description: as for outcome 3
Time Frame: as for outcome 3
Population: ITT population included all participants who were enrolled into the study.
Measure: Mean (Standard Deviation); unit: liter per hour (l/hr)
Arm/Group | Phase I Dose Escalation (250mg) | Phase I Dose Escalation (500mg) | Phase I Dose Escalation (750mg) | Phase I Dose Escalation (1000mg)
Number analyzed (Participants) | 6 | 9 | 6 | 12
liter per hour (l/hr)
  Fasted | 4288.456 (1319.322) | 5440.949 (4844.515) | 1518.748 (822.714) | 2649.954 (4617.049)
  Fed | 529.606 (99.532) | 391.046 (99.118) | 246.643 (72.970) | 231.383 (97.746)

9. Secondary Outcome: Phase 1: Volume of Distribution (Vz_F_obs) of Abiraterone Acetate
Description: Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired blood concentration of a drug. Volume of distribution is normally calculated by using equation volume of distribution =dose/initial concentration. Blood samples for pharmacokinetic (PK) measurements was taken on Day -7 at hour 0 (predose), at hours 1, 2, 4, 6, 8, and 12 (postdose). On Day -6 at 24 hour (postdose) and Day -5 at 48 hour (postdose). On Days 1, 8, 15, 22 of Cycle 1 and Day 1 of Cycles 2 and 3 (Predose).
Time Frame: as for outcome 3
Population: ITT population included all participants who were enrolled into the study.
Measure: Mean (Standard Deviation); unit: Liter (L)
Arm/Group | Phase I Dose Escalation (250mg) | Phase I Dose Escalation (500mg) | Phase I Dose Escalation (750mg) | Phase I Dose Escalation (1000mg)
Number analyzed (Participants) | 6 | 9 | 6 | 12
Liter (L)
  Fasted | 653.745 (447.316) | 10252.077 (12268.787) | 13688.367 (4265.429) | 25494.398 (18670.215)
  Fed | 3940.400 (1275.408) | 3418.280 (1934.384) | 2739.655 (1084.694) | 4068.885 (1462.613)

10. Secondary Outcome: Phase 2: Radiographic Progression Free Survival (RAD-PFS)
Description: RAD-PFS is the time interval from the date of first dose of abiraterone acetate therapy to the date of death or radiographic disease progression according to the RECIST (Response Evaluation Criteria In Solid Tumors) criteria. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: Up to 12 weeks from start of treatment
Population: ITT population included all participants who were enrolled into the study. RAD-PFS was not analyzed because of insufficient data to provide a meaningful estimate of the median and associated confidence interval (CI)
Measure: Median (Full Range); unit: days
Arm/Group | Phase II Dose Treatment
Number analyzed (Participants) | 13
days | NA [NA to NA] — The median survival is not reached and the confidence interval was not estimable

11. Secondary Outcome: Phase 2: PSA Progression Free Survival (PSA-PFS)
Description: PSA-PFS is the time interval from the date of first dose of abiraterone acetate therapy to the date of death or the PSA progression as defined by the Prostate Specific Antigen Working Group (PSAWG) criteria.
Time Frame: Up to 12 weeks from start of treatment
Population: ITT population included all participants who were enrolled into the study.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Phase II Dose Treatment
Number analyzed (Participants) | 33
days | 473 [281 to NA] — The median survival is not reached and the confidence interval was not estimable.

12. Secondary Outcome: Phase 2: Radiographic Objective Response Rate (RAD-ORR)
Description: The objective response rate is defined as the proportion of participants with measurable lesions achieving a Complete Response (CR) or Partial Response (PR) based on Response Evaluation Criteria In Solid Tumors (RECIST) criteria. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: Up to 12 weeks from start of treatment
Population: Thirteen evaluable participants with measurable disease at baseline were evaluated for radiographic objective response rate.
Measure: Number; unit: participants
Arm/Group | Phase II Dose Treatment
Number analyzed (Participants) | 13
participants
  Confirmed | 9 [38.6 to 90.9]
  Not Confirmed | 1 [0.2 to 36.0]

13. Secondary Outcome: Phase 2: Time to PSA Progression
Description: The time interval from the date of first dose of abiraterone acetate therapy to the date of the PSA progression as defined by the PSAWG criteria.
Time Frame: Up to 12 weeks from start of treatment
Population: ITT population included all participants who were enrolled into the study.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Phase II Dose Treatment
Number analyzed (Participants) | 33
days | 497 [281 to NA] — The median survival is not reached and the confidence interval was not estimable

14. Secondary Outcome: Phase 2: Duration of PSA Response
Description: Duration of PSA response was defined as the duration between the date of confirmed PSA response and subsequent PSA progression date as defined by the PSAWG criteria.
Time Frame: Up to 12 weeks from start of treatment
Population: ITT population included all participants who were enrolled into the study.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Phase II Dose Treatment
Number analyzed (Participants) | 33
days | 477 [283 to NA] — The median survival is not reached and the confidence interval was not estimable.

15. Secondary Outcome: Phase 2: Participants With Change in Eastern Cooperative Oncology Group (ECOG) Performance Status Score
Description: ECOG performance status score ranges from 0 to 5 where 0=fully active, perform all pre-disease activities without restriction. 1=restricted in physically strenuous activity but ambulatory, carry out work of a light or sedentary nature. 2=ambulatory, capable of self-care, unable to carry out any work activities, up and about more than (>) 50% of waking hours. 3=capable of limited self-care, confined to bed or chair >50% of waking hours. 4=completely disabled, not capable of any self-care, totally confined to bed or chair. 5=dead.
Time Frame: Up to 12 weeks from start of treatment
Population: ITT population included all participants who were enrolled into the study.
Measure: Number; unit: participants
Arm/Group | Phase II Dose Treatment
Number analyzed (Participants) | 33
participants
  Baseline ECOG 0 | 20
  Baseline ECOG 1 | 13
  Baseline ECOG 2 | 0
  Baseline ECOG 3 | 0
  Baseline ECOG 4 | 0
  Best Post-Baseline ECOG 0 | 28
  Best Post-Baseline ECOG 1 | 5
  Best Post-Baseline ECOG 2 | 0
  Best Post-Baseline ECOG 3 | 0
  Best Post-Baseline ECOG 4 | 0

16. Secondary Outcome: Phase 2: Overall Survival
Description: Overall survival is the time interval from the date of first dose (cycle 1 day 1) of abiraterone acetate therapy to the date of death from any cause.
Time Frame: Up to Month 60
Population: ITT population included all participants who were enrolled into the study.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Phase II Dose Treatment
Number analyzed (Participants) | 33
days | NA [NA to NA] — The median survival is not reached and the confidence interval was not estimable.

17. Secondary Outcome: Phase 2: Duration of Objective Response
Description: Duration of objective response was assessed only in participants who achieved a CR or PR, and measured from the first documented date of response to the first documented date of disease progression according to the RECIST criteria. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: Up to 12 weeks from start of treatment
Population: Thirteen evaluable participants with measurable disease at baseline were evaluated for radiographic duration of objective response.
Measure: Median (95% Confidence Interval); unit: days
Groups:
- Phase II Dose Treatment: The first cohort was a abiraterone acetate 250 mg/day orally (by mouth), once daily for 28-day treatment periods , if no dose limiting toxicity (DLT) was documented at this dose, the dose will be escalated to next dose levels 500, 750, and 1000 mg/day. The dose escalation will continue to a maximum of 1000 mg/day until maximum tolerated dose (MTD) and a recommended Phase II dose was established.
Arm/Group | Phase II Dose Treatment
Number analyzed (Participants) | 13
days | NA [253 to NA] — The median survival is not reached and the confidence interval was not estimable.

ADVERSE EVENTS:
Arm/Group | Phase 1 250 MG/DAY | Phase 1 500 MG/DAY | Phase 1 750 MG/DAY | Phase 1 1000 MG/DAY | Phase 2 1000 MG/DAY
Serious Adverse Events (participants affected / at risk) | 1/6 | 2/9 | 0/6 | 0/12 | 10/33
Other Adverse Events (participants affected / at risk) | 6/6 | 9/9 | 6/6 | 12/12 | 33/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1 250 MG/DAY (N=6) | Phase 1 500 MG/DAY (N=9) | Phase 1 750 MG/DAY (N=6) | Phase 1 1000 MG/DAY (N=12) | Phase 2 1000 MG/DAY (N=33)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Arrhythmia Supraventricular (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Myocardial Infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Ventricular Extrasystoles (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Oedema Peripheral (General disorders) | 0 | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 1
Cystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Device Related Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Urinary Tract Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 2
Urosepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 2
Troponin Increased (Investigations) | 0 | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 1
Pathological Fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 1 | 1 | 0 | 0 | 1
Calculus Bladder (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 2
Renal Failure (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Urinary Bladder Haemorrhage (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Urinary Incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Urinary Retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1 250 MG/DAY (N=6) | Phase 1 500 MG/DAY (N=9) | Phase 1 750 MG/DAY (N=6) | Phase 1 1000 MG/DAY (N=12) | Phase 2 1000 MG/DAY (N=33)
Lymphopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 2
Atrial Fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1 | 1
Palpitations (Cardiac disorders) | 0 | 1 | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Cerumen Impaction (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0
Hypoacusis (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 2
Adrenal Insufficiency (Endocrine disorders) | 0 | 1 | 0 | 1 | 0
Gynaecomastia (Endocrine disorders) | 0 | 0 | 0 | 1 | 3
Cataract (Eye disorders) | 1 | 0 | 0 | 1 | 1
Ocular Discomfort (Eye disorders) | 0 | 1 | 0 | 0 | 0
Ocular Hyperaemia (Eye disorders) | 0 | 1 | 0 | 1 | 0
Visual Acuity Reduced (Eye disorders) | 0 | 0 | 1 | 0 | 0
Abdominal Discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 2
Abdominal Distension (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 1 | 2 | 2 | 2 | 3
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2
Constipation (Gastrointestinal disorders) | 0 | 3 | 2 | 2 | 7
Defaecation Urgency (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 4 | 3 | 4 | 7
Dry Mouth (Gastrointestinal disorders) | 0 | 2 | 2 | 1 | 2
Dyspepsia (Gastrointestinal disorders) | 0 | 3 | 2 | 0 | 1
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Gingival Pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2
Lip Dry (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 3 | 1 | 6 | 5
Rectal Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 3
Vomiting (Gastrointestinal disorders) | 0 | 1 | 1 | 3 | 7
Asthenia (General disorders) | 1 | 3 | 2 | 2 | 2
Chills (General disorders) | 0 | 0 | 1 | 1 | 0
Fatigue (General disorders) | 3 | 7 | 4 | 8 | 16
Irritability (General disorders) | 1 | 0 | 1 | 0 | 0
Mucosal Dryness (General disorders) | 0 | 0 | 1 | 0 | 0
Oedema (General disorders) | 0 | 1 | 0 | 0 | 0
Oedema Peripheral (General disorders) | 1 | 4 | 0 | 6 | 9
Pain (General disorders) | 0 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 1 | 1 | 1
Tenderness (General disorders) | 0 | 0 | 0 | 1 | 0
Thirst (General disorders) | 0 | 1 | 0 | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 5
Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 3
Influenza (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Lower Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Tinea Versicolour (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 1 | 1 | 1 | 1 | 5
Urinary Tract Infection (Infections and infestations) | 0 | 0 | 0 | 2 | 3
Contrast Media Reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 2
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 3 | 5
Excoriation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 3
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 2
Joint Sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Muscle Injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Rib Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Skin Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 2
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Alanine Aminotransferase Increased (Investigations) | 0 | 0 | 1 | 0 | 4
Aspartate Aminotransferase Increased (Investigations) | 1 | 0 | 0 | 2 | 3
Blood Alkaline Phosphatase Increased (Investigations) | 1 | 0 | 1 | 1 | 2
Blood Bicarbonate Decreased (Investigations) | 0 | 0 | 0 | 1 | 0
Blood Creatinine Increased (Investigations) | 0 | 0 | 0 | 1 | 1
Platelet Count Decreased (Investigations) | 0 | 1 | 0 | 0 | 1
Weight Decreased (Investigations) | 1 | 0 | 0 | 0 | 2
Weight Increased (Investigations) | 0 | 0 | 0 | 1 | 0
White Blood Cell Count Decreased (Investigations) | 0 | 1 | 0 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 1 | 2 | 1 | 3 | 1
Decreased Appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 3
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 2 | 0 | 0
Hyperchloraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 2 | 5
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 2
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 2 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 3
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 4 | 4 | 10
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 5
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2 | 2 | 9
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 2 | 8
Bone Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 10
Flank Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1
Hypercreatinaemia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Muscle Fatigue (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 6
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 2 | 1 | 2 | 0 | 2
Musculoskeletal Discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 1
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 4
Rotator Cuff Syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 2
Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Aphasia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Ataxia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 2 | 3 | 7
Dizziness Postural (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 3 | 2 | 7 | 3
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Peripheral Sensory Neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 2
Transient Ischaemic Attack (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 0 | 0 | 1
Confusional State (Psychiatric disorders) | 0 | 0 | 0 | 1 | 2
Depressed Mood (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Depression (Psychiatric disorders) | 1 | 1 | 1 | 0 | 3
Euphoric Mood (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 1 | 0 | 0 | 3
Mood Altered (Psychiatric disorders) | 0 | 0 | 1 | 0 | 2
Personality Change (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Stress (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 1 | 1 | 0 | 1 | 2
Micturition Urgency (Renal and urinary disorders) | 0 | 0 | 1 | 1 | 0
Nocturia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 3
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 1 | 2 | 0
Urinary Incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 3
Urinary Retention (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 2
Urinary Tract Obstruction (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 1
Pelvic Pain (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0
Testicular Pain (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 4 | 1 | 5
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 0 | 2
Pharyngolaryngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Postnasal Drip (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1
Rales (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 2
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Actinic Keratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Dry Skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 8
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 4
Skin Hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 0
Hot Flush (Vascular disorders) | 0 | 2 | 2 | 3 | 10
Hypertension (Vascular disorders) | 2 | 2 | 3 | 5 | 7
Hypotension (Vascular disorders) | 1 | 2 | 0 | 0 | 3
Orthostatic Hypotension (Vascular disorders) | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days